CLINICAL TRIAL: NCT05780710
Title: Multicentric Prospective Clinical Study to Evaluate the Aktiia Optical Blood Pressure Monitoring (OBPM) Device Compared to Standard Home Blood Pressure Monitoring (HBPM) in Hypertensive Patients When Blood Pressure Lowering Medications Intake
Brief Title: OBPM_Meds2023: Multicentric Prospective Clinical Study to Evaluate the Aktiia Optical Blood Pressure Monitoring (OBPM) Device Compared to Standard Home Blood Pressure Monitoring (HBPM) in Hypertensive Patients When Blood Pressure Lowering Medications Intake
Acronym: OBPM_Meds2023
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OBPM_Meds2023
Record Dates: First submitted 2023-02-10; First posted 2023-03-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Intervention Model Description: Study participants are asked to wear the Aktiia bracelet continuously every day for 4 to 19 weeks in total, depending on the study group, and initialize their Aktiia bracelet with the Aktiia cuff at different timepoints.
  In parallel, GROUP 1 and 2 participants are asked to take 3 successive Blood Pressure lowering medications during 2 weeks per treatment. Treatment periods are followed by 2 weeks of washout. The order of drug intake is randomly assigned for every participant. GROUP 3 participants will receive and individualized antihypertensive medication assigned by the investigator.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meds2023 GROUP 1 (Other): GROUP 1 participants are asked to wear the Aktiia bracelet continuously every day for 13 weeks in total and initialize their Aktiia bracelet with the Aktiia cuff at different timepoints.
  In parallel, GROUP 1 participants are asked to take 3 successive Blood Pressure lowering drugs during 2 weeks per treatment. Treatment periods are followed by 2 weeks of washout (no treatment).
  Interventions: Other: Aktiia Optical Blood Pressure Monitoring (OBPM) device and antihypertensive drugs (monotherapy and bitherapy)
- Meds2023 GROUP 2 (Other): GROUP 2 participants are asked to wear the Aktiia bracelet continuously every day for 19 weeks in total and initialize their Aktiia bracelet with the Aktiia cuff at different timepoints.
  In parallel, GROUP 2 participants are asked to stop their previous antihypertensive monotherapy for the first 2 weeks of the study participation and then take 3 successive blood pressure-lowering medications during 2 weeks per treatment. Treatment periods are followed by 2 weeks of washout (no treatment). Finally, they resume their initial monotherapy intake for a period of 4 weeks.
  Interventions: Other: Aktiia Optical Blood Pressure Monitoring (OBPM) device and antihypertensive drugs (monotherapy)
- Meds2023 GROUP 3 (Other): GROUP 3 participants are asked to wear the Aktiia bracelet continuously every day for 4 weeks in total and initialize their Aktiia bracelet with the Aktiia cuff at different timepoints.
  In parallel, GROUP 3 participants are asked to take their initial antihypertensive medication that doesn't allow them to have controlled blood pressure for 1 week. For the following 3 weeks of the study participation, GROUP 3 participants are asked to take an individualized antihypertensive therapy assigned by the investigator.
  Interventions: Other: Aktiia Optical Blood Pressure Monitoring (OBPM) device and individualized antihypertensive treatment

INTERVENTIONS:
Other: Aktiia Optical Blood Pressure Monitoring (OBPM) device and antihypertensive drugs (monotherapy and bitherapy) — The device under test is Aktiia Optical Blood Pressure Monitoring (OBPM) device and the comparator is the Aktiia cuff.
  For study GROUP 1:
  Study drugs are:
  * Perindopril MEPHA (Angiotensin Converting Enzyme (ACE) inhibitors).
  * Indapamide MEPHA (Diuretics).
  * Amlodipine MEPHA (Calcium channel blockers). In each study treatment period, subjects in GROUP 1 will receive one of the following for each treatment period: monotherapy with Indapamide, bitherapy with Indapamide plus Perindopril, or bitherapy with Perindopril plus Amlodipine.
  Other Names: Aktiia system, Aktiia device, Aktiia bracelet, Aktiia cuff
  Arms: Meds2023 GROUP 1
Other: Aktiia Optical Blood Pressure Monitoring (OBPM) device and antihypertensive drugs (monotherapy) — Study drugs:
  * Perindopril MEPHA (Angiotensin Converting Enzyme (ACE) inhibitors).
  * Indapamide MEPHA (Diuretics).
  * Amlodipine MEPHA (Calcium channel blockers). In each study treatment period, subjects in GROUP 2 will receive one of the following monotherapies: Perindopril , Indapamide, or Amlodipine.
  Other Names: Aktiia system, Aktiia device, Aktiia bracelet, Aktiia cuff
  Arms: Meds2023 GROUP 2
Other: Aktiia Optical Blood Pressure Monitoring (OBPM) device and individualized antihypertensive treatment — For study GROUP 3:
  Subjects will be prescribed an individualized new antihypertensive treatment at their consultation with the Investigator at Visit 1.
  Other Names: Aktiia system, Aktiia device, Aktiia bracelet, Aktiia cuff
  Arms: Meds2023 GROUP 3

SUMMARY:
Study design: Prospective, multicentric, randomized, comparative study Study duration: between 4 and 19 weeks depending on the study group. Population: minimum 35 hypertensives (stage 1 or stage 2) participants divided into 3 groups depending on hypertension criteria. GROUP 1 = untreated hypertensives, stage 1 or stage 2; GROUP 2 = hypertensives, stage 1, who are taking antihypertensive monotherapy; GROUP 3 = hypertensives, stage 1 or stage 2, who are taking antihypertensive treatment that doesn't allow them to have controlled blood pressure.

Device Under Test (DUT): Aktiia device Reference: HBPM (Aktiia cuff) Periods of treatment: For GROUPS 1 and 2, 2 weeks of treatment for each antihypertensive medication followed by a washout period of 2 weeks (3 antihypertensive medications in total with a fixed dose; medication intake order is randomly assigned). For GROUP 3, an individualized new antihypertensive medication will be prescribed during the consultation with the investigator that will be administered for 3 weeks.

DETAILED DESCRIPTION:
This study with N = 35 participants minimum, over 2 to 6 visits, depending on the study group, has been designed to compare Aktiia device systolic and diastolic blood pressure measurements against HBPM reference measurements in participants taking 3 successive BP-lowering medications during 2 weeks per treatment for GROUPS 1 and 2, while GROUP 3 will receive, during 3 weeks, an individualized medication decided by the investigator. For GROUPS 1 and 2, periods of treatment are followed by 2 weeks of washout.

Study participants are: For GROUP 1, hypertensive Stage 1 (SBP 140-159 mmHg or DBP 90-99 mmHg) or hypertensive Stage 2 (SBP 160-179 mmHg or DBP 100-109 mmHg) that are naive of antihypertensive treatments at the inclusion in the study. For GROUP 2, hypertensives Stage 1 (SBP 140-159 mmHg or DBP 90-99 mmHg) with no other cardiovascular risk factors who are taking an antihypertensive monotherapy, for whom previous treatment will be stopped at the study inclusion and will be resumed for the last 4 weeks of the study participation. For GROUP 3, uncontrolled hypertensive Stage 1 (SBP 140-159 mmHg or DBP 90-99 mmHg) or hypertensive Stage 2 (SBP 160-179 mmHg or DBP 100-109 mmHg) who are taking antihypertensive treatment that doesn't allow them to have controlled blood pressure.

Study participants are asked to:

Wear the Aktiia bracelet continuously every day for 4 to 19 weeks in total, depending on the study group, Initialize their bracelet with the Aktiia cuff at different time points, Measure their blood pressure with an HBPM (Aktiia cuff) twice per day, Take their BP-lowering medications during the treatment periods, Complete 2 to 3 different surveys, depending on the study group, to give their feedback on Aktiia product use compared to HBPM.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 21 to 85 years old
2. Subjects that can read and speak French
3. Subjects that own a smart phone that uses either the iOS or Android operating system
4. Hypertensive Stage 1 (SBP 140-159 mmHg or DBP 90-99 mmHg) or Hypertensive Stage 2 (SBP 160-179 mmHg or DBP 100-109 mmHg) or for subjects aged > 65yo SBP ≥160 mmHg,
5. Naive of antihypertensive drugs at the inclusion in the study (no antihypertensive drugs taken in the last 3 months before Visit 1) and during the conduct of the study apart from the study drugs
6. Subjects agreeing to attend all 4 on-site visits and follow study procedures
7. Subjects that have signed the informed consent form

Exclusion Criteria:

1. Subjects have contraindications to the study drugs
2. Subjects with Hypertension Stage 3 (SBP/DBP >180/110 mmHg)
3. Subjects with orthostatic hypotension (a 20 mmHg decrease in systolic BP, or 10 mmHg decrease in diastolic BP when measured in the standing position after a 1-minute waiting period)
4. Subjects who are likely to be unable to perform the HBPM required for the study within the designated time frame (7 to 11

   a.m. and 4 to 9 p.m.).
5. Subjects having medical interventions or taking treatments during the study that could have an impact on their BP
6. For GROUPS 1 and 2 only: Subjects with target organ damage (left ventricular hypertrophy observed on ECG, and/ or, albumin/creatinine ratio in urine ≥3.5 mg/mmol)
7. Subjects with tachycardia (heart rate at rest > 120bpm)
8. Subjects with atrial fibrillation
9. Cardio myopathy (FE<40%)
10. Severe valvular disease
11. Implanted devices such as a pacemaker or defibrillator
12. Subjects with diabetes
13. Subjects with renal dysfunctions (eGFR < 45mL/min/1.73 m2 for patients between 21-85 yo)
14. Subjects with hyper-/hypothyroidism
15. Subjects with pheochromocytoma
16. Subjects with Raynaud's disease
17. Subjects with an arteriovenous fistula
18. Women in known pregnancy
19. Subjects with trembling and shivering
20. Subjects with lymphoedema
21. Low or elevated potassium level: threshold ≤3.5 mmol/L or ≥4.8 mmol/L
22. Presence of an intravascular device
23. Subjects with exfoliative skin diseases
24. Subjects with arm paralysis
25. Subjects with arm amputation
26. Subjects with upper arm circumference < 22cm or > 42cm
27. Subjects with wrist circumference > 23cm
28. Subjects with non-standard circadian rhythm, including shift workers and night workers
29. Subjects who have received a mastectomy.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Daytime Systolic and Diastolic Blood Pressure averages (last 3 days of week 1 versus last 3 days of week 3) | Last 3 days of the washout period (week 1), against the last 3 days of the treatment period (week 3)
  Statistics on the comparison of the changes in average daytime Blood Pressure values pre- and post-intervention between the two modalities (Aktiia device and HBPM)
Daytime Systolic and Diastolic Blood Pressure averages (last 3 days of week 5 versus last 3 days of week 7) | Last 3 days of the washout period (week 5), against the last 3 days of the treatment period (week 7)
  Statistics on the comparison of the changes in average daytime Blood Pressure values pre- and post-intervention between the two modalities (Aktiia device and HBPM)
Daytime Systolic and Diastolic Blood Pressure averages (last 3 days of week 9 versus last 3 days of week 11) | Last 3 days of the washout period (week 9), against the last 3 days of the treatment period (week 11)
  Statistics on the comparison of the changes in average daytime Blood Pressure values pre- and post-intervention between the two modalities (Aktiia device and HBPM)

SECONDARY OUTCOMES:
Participant's compliance | GROUP 1= 13 weeks; GROUP 2= 19 weeks; GROUP 3= 4 weeks.
  Number of measurements made each day by the Aktiia System
Participant's compliance | GROUP 1= 13 weeks; GROUP 2= 19 weeks; GROUP 3= 4 weeks.
  Number of successful synchronizations with the Aktiia System
Participant's perception | GROUP 1= 13 weeks; GROUP 2= 19 weeks; GROUP 3= 4 weeks.
  Compilation of answers to the surveys

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - HUG, Geneva, Canton of Geneva
  - CHVR, Sion, Valais
  - CHUV, Lausanne